CLINICAL TRIAL: NCT01083329
Title: Effect of Nicotinic Acid on Adipose Tissue Inflammation in Obese Subjects
Acronym: ANITA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0816302
Record Dates: First submitted 2010-02-25; First posted 2010-03-09 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Obesity
Keywords: nicotinic acid; lipolysis; training program; adipose tissue inflammation; obese
MeSH Terms: conditions — Obesity | interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): for 16 weeks
  Interventions: Behavioral: training; Drug: Placebo
- nicotinic acid (Active Comparator): for 16 weeks :
  * week 1 = 375 mg per day,
  * week 2 = 500 mg per day,
  * week 3 = 750 mg per day,
  * week 4 = 1000 mg per day,
  * week 5 = 1500 mg per day,
  * weeks 6 to 16 = 2000 mg per day.
  Interventions: Behavioral: training; Drug: nicotinic acid

INTERVENTIONS:
Behavioral: training — the last 8 weeks, the subjects will follow a training program calculated to optimize use of lipid
Drug: nicotinic acid — Obese subjects will receive nicotinic acid or placebo for 16 weeks
  Arms: nicotinic acid
Drug: Placebo — Obese subjects will receive nicotinic acid or placebo for 16 weeks
  Arms: placebo

SUMMARY:
Our working hypothesis postulates that lipolysis is a determinant of inflammation in adipose tissue (AT). Inhibition of lipolysis, e.g. using the oldest normolipidemic drug, nicotinic acid, has proved valuable to combat the metabolic syndrome. Our proposal will determine whether part of the beneficial effects of this antilipolytic compound is due to a diminution of AT inflammation.

To this aim, the effect of nicotinic acid or placebo will be studied in male obese subjects with or without a training program which goal is to enhance lipolysis.

DETAILED DESCRIPTION:
24 male obese insulin resistant subjects will receive nicotinic acid or placebo for 16 weeks. The last 8 weeks, the subjects will follow a training program calculated to optimize use of lipid. Insulin sensitivity and glucose tolerance will be assessed using, respectively, fasting-based estimates of insulin sensitivity (plasma and muscle) and oral glucose tolerance test. Plasma parameters of adipokines and, inflammatory and metabolic parameters will be determined. As an index of AT inflammation, the percentage and the phenotype of macrophages will be determined using flow cytometry of cells of the stromavascular fraction of subcutaneous AT. Macrophage infiltration will be investigated by light microscopy. The characterization of the inflammatory profile of AT will be completed by measurements of the expression of genes that are either specific markers of human AT macrophages or inflammatory and anti-inflammatory adipokines. This combination of approaches has never been carried out during a pharmacological intervention in humans. The following points will be addressed:

* determine the influence of lipolysis on AT inflammation, specifically on macrophage activation and adipokine production.
* examine the causal relationship between adipocyte FA metabolism, AT inflammation and insulin sensitivity.
* establish whether the beneficial effect of antilipolytic drugs may be attributable at least in part to a decrease in AT inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent form
* Age 25 to 45 year-old
* Male, insulin resistant obese subjects (30<BMI<40 kg/m2),
* Blood arterial pressure<140/90 mmHg

Exclusion Criteria:

* History of cardiovascular disease
* Treatment with drugs which can interfere with cardiovascular system and autonomic nervous system (i.e. beta blockers).
* Treatment with nicotinic acid
* Treatment with fibrates, statins, cholestyramine and ezetimibe
* Treatment with thiazidics
* Fasted hyperglycaemia > 1,26 g/l (Diabetes)
* Triglycerides >5 g/l
* Blood arterial pressure > 140/90 mm Hg

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Comparison of changes of AT inflammation will be measured by gene expression analysis | Visit 1(T0), Visit 2 (T+8 weeks of treatment) and Visit 3 (T+16 weeks of treatment)

SECONDARY OUTCOMES:
Comparison of changes in insulin sensitivity and glucose tolerance | Visit 1(T0), Visit 2 (T+8 weeks of treatment) and Visit 3 (T+16 weeks of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Thalamas, Principal Investigator — University Toulouse Hospital
Locations (1):
- Centre d'Investigation Clinique, Purpan University Toulouse Hospital, Toulouse, France

REFERENCES:
- [Result] Montastier E, Beuzelin D, Martins F, Mir L, Marques MA, Thalamas C, Iacovoni J, Langin D, Viguerie N. Niacin induces miR-502-3p expression which impairs insulin sensitivity in human adipocytes. Int J Obes (Lond). 2019 Jul;43(7):1485-1490. doi: 10.1038/s41366-018-0260-5. Epub 2018 Nov 27. PMID 30482933
- [Derived] Bourlier V, Saint-Laurent C, Louche K, Badin PM, Thalamas C, de Glisezinski I, Langin D, Sengenes C, Moro C. Enhanced glucose metabolism is preserved in cultured primary myotubes from obese donors in response to exercise training. J Clin Endocrinol Metab. 2013 Sep;98(9):3739-47. doi: 10.1210/jc.2013-1727. Epub 2013 Jul 24. PMID 23884778